CLINICAL TRIAL: NCT01253278
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Effects of Multiple Escalating Oral Doses of LY2393910 in Patients With Type 2 Diabetes Mellitus
Brief Title: A Multiple-Ascending Dose Study in Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 13183; I4B-FW-GPCB (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 20 mg LY2393910 (Experimental)
  Interventions: Drug: LY2393910
- 60 mg LY2393910 (Experimental)
  Interventions: Drug: LY2393910
- 150 mg LY2393910 (Experimental)
  Interventions: Drug: LY2393910
- 450 mg LY2393910 (Experimental)
  Interventions: Drug: LY2393910
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2393910 — as capsules, administered orally once daily for two weeks
  Arms: 150 mg LY2393910; 20 mg LY2393910; 450 mg LY2393910; 60 mg LY2393910
Drug: Placebo — as capsules, administered orally once daily for two weeks
  Arms: Placebo

SUMMARY:
The study drug LY2393910 is being evaluated as a possible treatment for diabetes. The primary purpose of a patient's participation in this study is to help answer the following research question(s), and not to provide treatment for diabetes:

* The safety of LY2393910 and any side effects that might be associated with it following 2 weeks of doses
* How long it takes the body to absorb and remove LY2393910 following dosing over 2 weeks
* How daily dosing of LY2393910 affects blood levels of sugar (glucose), insulin and other naturally occurring substances in your body
* How daily dosing of LY2393910 affects the cells that produce insulin
* Any differences in the above between LY2393910 taken as daily doses in the morning or in the evening

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus
* Must be on a stable treatment regimen (maintained on diet/exercise therapy with or without metformin) for at least 4 weeks prior to study entry
* Have a glycated haemoglobin (HbA1c) value greater than or equal to 6.5% and less than or equal to 10.0% on a stable treatment regimen
* Weigh 45.0 kg or more
* Have a Body Mass Index (BMI) greater than or equal to 18.5 and less than or equal to 40.0 kg/m2
* Are willing and able to conduct self-blood glucose monitoring tests

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days from a clinical trial involving use of an investigational drug or device other than the study drug used in this study, or are concurrently enrolled in any other type of medical research judged not to be compatible with this study
* Use of insulin for diabetic control for more than 6 consecutive days within 1 year prior to study entry
* Use of thiazolidinediones within 3 months, or other oral anti-diabetics (OADs), apart from metformin, within 1 month prior to study entry. Metformin is acceptable for this study
* Previous myocardial infarction, stroke or transient ischaemic event ('TIA'), or clinically significant coronary events or symptoms within 6 months prior to study entry
* Subjects who have any evidence of heart insufficiency, hypokalaemia, family history of long-QT-syndrome or are receiving other drugs which extend the QT interval
* Clinically significant peripheral vascular disease
* Clinical evidence of active diabetic proliferative retinopathy
* Known significant autonomic neuropathy
* Any patient having experienced a keto-acidotic episode requiring hospitalisation in the last 6 months
* Symptomatic hyperglycemia exhibited by significant osmotic symptoms (polyuria or polydipsia), unanticipated weight loss or dehydration
* Evidence of hepatitis B and/or positive hepatitis B surface antigen, at screening
* Subjects who have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females)
* Subjects who are heavy smokers (> 10 cigarettes, or equivalent, per day) or are unable or unwilling to refrain from nicotine during CRU admissions

Exclusion Criteria for EU Site only --

* Regular use of known drugs of abuse and/or positive findings on urinary drug screening
* Evidence of human immunodeficiency virus (HIV) and/or positive HIV antibodies
* Evidence of hepatitis C and/or positive hepatitis C antibodies

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Clinically Significant Effects | Over four weeks

SECONDARY OUTCOMES:
Pharmacokinetics of LY2393910, Area Under the Curve (AUC) | From predose Day 1 up until Day 19
Change from baseline to day 28 in glucagon | Baseline, day 28
Pharmacokinetics of LY2393910, maximum concentration (Cmax) | From predose Day 1 up until Day 19
Change from baseline to day 28 in glucose-like peptide 1 (GLP-1) | Baseline, day 28
Change from baseline to day 14 in insulin | baseline, day 14
Change from baseline to day 14 in proinsulin | baseline, day 14
Change from baseline to day 28 in glucose | baseline, day 28
Change from baseline to day 14 in C-peptide | baseline, day 14

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neuss, Germany